CLINICAL TRIAL: NCT00451503
Title: Evaluation of Middle Ear Implants in the Therapeutic Strategy of Auditory Rehabilitation in Case of Failure of Conventional Hearing Aid
Brief Title: Evaluation of Middle Ear Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P051023
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Hearing Loss
Keywords: Hearing; Auditory rehabilitation; Middle ear implant; Surgery
MeSH Terms: conditions — Hearing Loss | interventions — Ossicular Prosthesis; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): surgery
  Interventions: Device: Middle Ear Implant

INTERVENTIONS:
Device: Middle Ear Implant — surgery
  Other Names: surgery

SUMMARY:
The middle ear implant are used for patients with mild to severe sensorineural hearing loss, who cannot benefit from conventional hearing aids because of medical reasons such as chronic external otitis or external skin irritation. The device is also available for patients who are dissatisfied with the conventional hearing aids because of poor sound quality, feedback or occlusion of the ear canal. To date, more than 1500 patients have been implanted in Europe and about more than 600 patients in France. The aim of the present study is to compare in a randomized study the performances of the system to those of the conventional hearing aid in patients with similar degree of hearing loss.

DETAILED DESCRIPTION:
Objective: The main objective of this study is to demonstrate that the middle ear implant increases the hearing in terms of speech intelligibility in quiet and noisy conditions, in patients who have no further benefit of their conventional hearing aid. The quality of life of these patients will be evaluated as well as the tolerance of the middle ear implant after 6 months.

Design of the study: 420 patients with mid or severe hearing loss will be included. They will have for 3 months the best conventional hearing aid adapted to their hearing loss. The first 84 patients who will not have a benefit of this hearing aid, will be randomised in two groups. The patients of the first group will be operated as soon as possible, the surgery of the patients of the second group will be delayed by 6 months. The whole duration of the study is 48 months.

Evaluation criteria: Audiological testing (pure-tone hearing thresholds, speech comprehension in quiet and noise), and subjective evaluation using self-assessment scales will be performed before and 6 months after the implantation in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adults patients
* hearing loss
* accept to participate
* having health insurance

Exclusion Criteria:

* known disease that needs MRI follow up
* contraindication to middle ear surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-03; Primary Completion 2011-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the middle ear implant on speech intelligibility in quiet and noise in case of failure of conventional hearing aid | during the study

SECONDARY OUTCOMES:
Assessment of the life quality of patients | during the study
Assessment of the tolerance at 6 months postoperative of the middle ear | 6 months postoperative
implantation | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Olivier STERKERS, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Beaujon, Clichy, France